CLINICAL TRIAL: NCT03736044
Title: Analysis of T Cell Population to Obtain a Free-drug Remission in Patients Affected by Rheumatoid Athritis in Remission Phase Induced by TNF-blocker Therapy
Brief Title: Reconstitution of CD4+CD25highCD127low/-Tcell
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital of Ferrara (Other)
Responsible Party: Principal Investigator, Andrea Lo Monaco, Rheumatology Physician assistant/Principal investigator, University Hospital of Ferrara
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PRUa1GR-2013 -00000156
Record Dates: First submitted 2018-10-11; First posted 2018-11-08 (Actual); Last update posted 2018-11-08 (Actual); Status verified 2018-11

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid arthritis; Remission; T regulatory lymphocytes; Tumor Necrosis Factor-blocker therapy
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Intervention Model Description: * Group A: patients on treatment with TNF-blockers plus DMARDs
  * Group B: patients treated with DMARDs only (Methotrexate/Leflunomide), never treated with anti-TNF.
  In addition a cohort of healthy subjects matched for sex and age used as a control.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TNF-blockers withdrawal (Experimental): Patients on treatment with TNF-blockers plus DMARDs in which a withdrawal of anti-TNF therapy was made.
  Interventions: Drug: TNF-blockers suspension in patients with rheumatoid arthritis
- DMARDs control group (No Intervention): Patients treated with DMARDs only (Methotrexate/Leflunomide), never treated with anti-TNF.

INTERVENTIONS:
Drug: TNF-blockers suspension in patients with rheumatoid arthritis — in patients treated with anti-TNF the intervention consisted in anti-TNF drug withdrawal, after a preliminary careful examination of remission status; a 18 months (at least) follow up was performed.
  Arms: TNF-blockers withdrawal

SUMMARY:
Rheumatoid arthritis (RA) is a systemic disabling inflammatory disease, of autoimmune origin characterized by chronic synovial inflammation resulting in joint damage. Treg cell function in patients with active RA is assumed to be impaired, a trend that seems to be reversed by TNFalpha antagonist therapy. Remission is the current treatment goal in RA.

An increasing number of patients in clinical trials achieve this goal raising the question whether patients who have been in remission for a prolonged period (sustained remission) still need medication indefinitely. From a decade TNF-blocker therapy have represented a new treatment option for RA patients non responders to conventional DMARDs and some evidence are now available showing that sustainable remission can be maintained achieved after withdrawal of TNF blocker. Objectives: to verify whether in RA patients in prolonged clinical and instrumental remission the percentages of CD4+CD25highCD127low/- T cells could represent a reliable marker of immunological remission and, even more relevant, if the pharmacological reconstitution of this "immune-modulator" Tcell population could contribute to better identify patients with a low risk of relapse after cessation of TNF-blocker therapy. Methods: in RA patients, who fulfilled the 1987 ACR revised criteria, with disease duration ! 5 years, clinical [Disease Activity Score on 28 joints-DAS28 0.56 ×√(TJC28) + 0.28×√(SJC28) + 0.70×ln(ESR) + 0.014×GH.TJC= Tender Joints Count (from 0 to 28); SJC= Swollen Joints Count (from 0 to 28) ESR=Erythrocyte Sedimentation Rate GH= patient's assessment of general health (VAS range from 0 to 100 mm); disease's flare was considered if: DAS44 >=2.4/DAS28 >=3.2.)], instrumental (joint ultrasonography: sites to be explored wrists are II-III metacarpophalangeal joint bilaterally using Power Doppler signal (grading 0-3); any other joint will be studied if symptomatic) and immunological (circulating CD4+CD25highCD127low/-Tcells and inflammatory cytokines levels) examination will be performed in order to asses, at different levels, disease activity status. Expected results: to identify in RA patients treated with anti-TNF an "exit-strategy" from these drugs based on clinical, imaging and immunologic features indicative of a sustained remission and to verify whether such conditions are able to predict a low incidence of relapse.

DETAILED DESCRIPTION:
1. To evaluate the incidence of disease flare after cessation of anti-TNF therapy in patients that meet sustained clinical and instrumental remission criteria together with reconstitution of the CD4+CD25highCD127low/- Tcell population respect to those patients in the same remission status with persistent low CD4+CD25highCD127low/- Tcell population.
2. Assessment of CD4+CD25highCD127low/- Tcell population behaviour induced by different drug treatments (anti-TNF vs DMARDs) in patient with RA who have achieved a prolonged remission status.
3. To assess the predictive value of modifications of CD4+CD25highCD127low/- Tcell population in patients who relapse.

Study design: all RA patients satisfying inclusion criteria will undergo to a baseline clinical, instrumental and immunologic evaluation. Peripheral CD4+CD25highCD127low/- Tcell population will be checked for and patients will be stratified in 2 groups:

* Group A: patients on treatment with TNF-blockers plus DMARDs
* Group B: patients treated with DMARDs only (Methotrexate/Leflunomide), never treated with anti-TNF In addition a cohort of healthy subjects matched for sex and age will be used as a control.

Patient's blood samples will be centralized at the "Laboratories of Technology for Advanced Therapies" of the University of Ferrara (www.ltta.tecnopoloferrara.it) directed by Prof. Paola Secchiero.

In group A anti-TNF drugs will be withdrawn and patients will be followed up. Patients belonging to the group B will be followed up without any further intervention. A tight clinical monitoring will be instituted and disease flares-up will be recorded. In case of disease flare therapeutic adjustment will be provided to the patients by the attending specialist team accordingly to the current standard of care.

ELIGIBILITY:
Inclusion Criteria:

* patients with RA fulfilling the 1987 ACR classification criteria (10) treated with anti-TNF and/or conventional DMARDs for at least 12 months, in prolonged remission (DAS28 <2.6 or DAS44 <1.6) for at least 6 months (checked in two consecutive visits 3 months apart), without Glucocorticosteroid (for at least 3 months, before), on a stable treatment for at least 3 months.

Exclusion Criteria:

* assumption of glucocorticosteroids within the three months before; confounding comorbidities such as fibromyalgia; chronic inflammatory disease other than RA; ongoing infections at the time of enrolment; recent trauma.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2013-11-25 (Actual); Primary Completion 2017-03-13 (Actual); Study Completion 2017-03-13 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects who flare-up after cessation of anti-TNF therapy after 24 months | 24 months
  disease flare-up defined as DAS 28 >3.2

SECONDARY OUTCOMES:
Proportion of subjects who are still in remission or il low disease activity after 3, 6, 9, 12, 15, 18, 21, 24 months | 24 months
  disease remission/low disease activity defined as DAS 28 <=3.2
Swollen joint counts after 3, 6, 9, 12, 15, 18, 21, 24 months | 24 months
  Number of Swollen Joints (range from 0 to 28) at clinical examination
Tender joint counts after 3, 6, 9, 12, 15, 18, 21, 24 months | 24 months
  Number of Tender joints (range from 0 to 28) at clinical examination
Patient self assessment of pain (VAS) after 3, 6, 9, 12, 15, 18, 21, 24 months | 24 months
  Severity of pain measured by visual analogic scale (0-10)
Physician's and patient's assessment of global disease activity (VAS) after 3, 6, 9, 12, 15, 18, 21, 24 months | 24 months
  Physician and Patient evaluation of Global disease activity measured by visual analogic scale (0-100)
HAQ (Health Assessment Questionnaire) after 3, 6, 9, 12, 15, 18, 21, 24 months | 24 months
  Evaluation of disability by HAQ. There are 8 sections: dressing, arising, eating, walking, hygiene, reach, grip, and activities. There are 2 or 3 questions for each section. Scoring within each section is from 0 (without any difficulty) to 3 (unable to do).The 8 scores of the 8 sections are summed and divided by 8.

IPD SHARING:
Plan to Share IPD: No